CLINICAL TRIAL: NCT06329362
Title: Quantitative Assessment of Bone Comparing the Minimally Invasive Ridge Splitting Versus the Conventional Open Flap Technique
Brief Title: Minimally Invasive Ridge Splitting Versus the Conventional Open Flap Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal College of Surgeons of Edinburgh (Other)
Responsible Party: Principal Investigator, Bassem Emad AbdElMoneim, Oral and Maxillofacial Surgeon, The Royal College of Surgeons of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-7-23
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Invasive Implant ridge splitting (Active Comparator): Using minimally invasive implant placement in atrophied ridge without mucoperiosteal flap, and specially designed implant shaped expanders.
  Interventions: Procedure: Minimally invasive implantation
- conventional open flap ridge splitting implantation. (Active Comparator): Using the conventional open flap technique with mucoperiosteal elevation to expose the ridge with the use of conventional bone expanders and chisels.
  Interventions: Procedure: Open flap procedure for ridge expansion.

INTERVENTIONS:
Procedure: Minimally invasive implantation — Specially designed ridge splitting instrumentation by Champions Implant GmbH which is implant shaped expanders.
  Other Names: Champions Implant GmbH
  Arms: Minimal Invasive Implant ridge splitting
Procedure: Open flap procedure for ridge expansion. — Mucoperiosteal elevation and ridge splitting using conventional ridge expanders.
  Other Names: Ridge splitting.
  Arms: conventional open flap ridge splitting implantation.

SUMMARY:
The goal of this clinical trial is to compare implant stability, and crestal bone loss, when using minimal invasive ridge splitting versus convenient open flap technique. The main question is Does Minimal Invasive Implant ridge splitting ("transmucosal" without flap) influence the implant stability and crystal bone loss, when compared with the conventional open flap techniques? Researchers will compare Group A: Minimal Invasive Implant ridge splitting and Group B: Triangular flap technique is used to see if there is significant difference between the two groups when measuring implant stability, and crestal bone density.

DETAILED DESCRIPTION:
Diagnostic stage:

Explanation of the operative procedure and obtaining the participants consent. Comprehensive clinical examination and understanding of participants chief complains and needs will be carried out.

CBCT acquisition:

Cone Beam Computed Tomography (CBCT) scans for the participants will be Taken preoperatively to determine the following:

1. Bone density (D1 & D4 for exclusion, while D2 & D3 shall be included)
2. To confirm the ridge mapping indicating alveolar ridge class IV. (Where height is adequate > 10mm, while width is "3-4 mm").

Planning the surgical procedure:

All planned surgical procedure will be carried out by main candidate under supervision.

Implant are planned to be placed (2 implants are placed in each segment "30-40 mm")

Surgical procedure:

Scrubbing and draping of the participants will be carried out in a standard fashion.

Local anesthesia (lidocaine 2%o,1/100000 adrenaline) Group A: Minimal Invasive Implant ridge splitting. A horizontal incision is made using fine end bur with high-speed hand piece deep from the edge of the ridge, passing down the cortical plate to the depth of the spongy bone, without mucoperiosteal elevation.

Using specially designed implant like bone expanders (Champions implants GmbH) to widen ridge with sequential application (which are 2.4, 2.8, 3.0, 3.3,3.8,4.3, and 5.3 mm in Diameter).

With each step the investigators shall carefully check the bone integrity and depth using calibrated probe.

By reaching the desired depth and width (till size 3.3 condensers and place 3.5 x 8 mm implants as a standard, using torque gage adjusted at 30-40 Newton's, that's to avoid pressure that might lead to initial resorption.

Closure of the incision line using interrupted suturing.

Group B: Triangular flap technique is used. With the horizontal component on the ridge and the vertical component posteriorly to avoid injury to the mental nerve, allowed by mucoperiosteal elevation to expose the target area.

2 vertical cuts on both ends to facilitate the ridge expansion, without the risk of crack or fracture of the buccal segment using conventional chisels till reaching the desired width that would accommodate the same implant diameter as for group A.

ELIGIBILITY:
Inclusion criteria:

1. Patients with atrophic posterior mandibular ridge with edentulous area 30-40 mm, minimum width 3-4 mm, and adequate height indicated for implant placement >9 mm.
2. Patient with Bone density D2 and D3.
3. Good general systemic condition.
4. Committed patient to attend follow up appointment.

Exclusion criteria:

1. Patients with systemic diseases that may affect the healing process of hard or soft tissues (e.g., uncontrolled diabetes mellitus).
2. Patient on medication that could hinder the normal healing process (e.g., steroids, immunosuppressant)
3. Patients with intra-bony lesions or infections.
4. Patient with bad habits (e.g. alcohol or Substance abuse).
5. Patient who received head and neck radiotherapy or chemotherapy in the last 10 years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Implant stability. | immediate postoperative, 1, 2, and 3 months post operative.
  Implant Stability Quotient (ISQ) evaluation via Ostell device for implant stability measurement, it measures on a scale from 1 to 100 and is a measure of the stability of an implant, less than 60 indicates low stability, 60-69 indicates medium stability, 70 and more indicates high stability.
  Method of aggregation: Mean and standard deviation.
  .
CBCT assessment | measurement points: preoperative, immediately postoperative, and 12 months postoperative, unless indicated otherwise e.g., Complications).
  Bone density at the implant site in House field unit. A Hounsfield unit reading of 1250 and above indicates D1 bone. A Hounsfield reading between 850 to 1250 units is indicative of D2 bone. A Hounsfield reading between 350 and 850 units is indicative of type D3 bone. A Hounsfield reading between 150 and 350 units is indicative of D4 bone. Method of aggregation: Mean and standard deviation.

SECONDARY OUTCOMES:
Postoperative Pain | to be completed by day 7 postoperative, describing the pain felt.
  Specific measurement variable: Visual Analogue Scale (VAS Scale), scale chart to be completed by the patient from 0-10 where 0 means no pain and 10 means worst of pain.
  Participant -level analysis: Final value. Method of aggregation: Mean and standard deviation
Operation Time | Time of the procedure from the beginning to the end.
  Specific measurement variable: operating time in minutes and seconds from the beginning to the end of the procedure.
  Participant-level analysis: Final value. Method of aggregation: Mean and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Emad Deif, Prof., Study Chair — Head of Oral and Maxillofacial Surgery Department - Faculty of Dentistry Cairo University
Locations (2):
- Faculty of Dentistry Cairo University, Cairo, Egypt
- Future Dental Academy GmbH, Flonheim, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No